CLINICAL TRIAL: NCT05081635
Title: Definitions of Success and Failure in Post-graduate Medical Education and Its Influencing Factors: A Delphi Consensus Study
Brief Title: Consenso2_F1 Delphi Consensus Study on Post-graduate Medical Education Success and Failure and Its Influencing Factors
Status: Completed | Type: Observational
Sponsor: Centro Hospitalar do Baixo Vouga (Other)
Collaborators: Conselho Nacional do Internato Médico (Unknown)
Responsible Party: Principal Investigator, Nuno Filipe Maio Lopes Fernandes, Principal Investigator, Centro Hospitalar do Baixo Vouga
Other Study IDs: Consenso2_Fase1
Record Dates: First submitted 2021-10-05; First posted 2021-10-18 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Medical Education

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Delphi panel: The Delphi panel will include 30 Portuguese experts in post-graduate medical education. The expert panel will include participants from the residency programs directors' coordination group, from the medical residents representing committee, from patients representing associations, from health institutions management teams, from the Portuguese Medical Association and also authors of relevant scientific articles on medical education. Study participants will be required to answer the questions of 3 questionnaires included in each of the 3 rounds of the study.

SUMMARY:
The objective of this study is to generate expert consensus statements on the definitions of success and failure and its influencing factors in Post-graduate medical education.

DETAILED DESCRIPTION:
A study will be performed using a e-Delphi process with Portuguese expert panel to generate recommendation statements related to the definitions of success and failure in Post-graduate medical education and its influencing factors and to determine the level of agreement for each statement from the panel as a whole. The following topics will be covered:

1. Success in Post-graduate medical education: definition, influencing factors
2. Failure in Post-graduate medical education: definition, influencing factors
3. Management Consensus is achieved through iterative rounds of survey and revision to the statements until a pre-determined level of agreement is met (75% agreement).

Part 1: planning and evidence review

* Series of planning sessions with study investigators
* Literature is reviewed/summarized
* Initial statements will be developed based on Round 1 results. Round 1 will be composed of 4 open-ended questions

Part 2: Survey to achieve consensus

* Survey, based on the initial statements developed on Round 1 results
* At least 2 additional rounds of review (remote rounds using an online platform) will be held to achieve consensus on each topic of interest and finalize consensus statements

ELIGIBILITY:
Inclusion Criteria:

* residency programs directors,
* members of the medical residents representing committee,
* members of patients representing associations,
* members of health institutions management teams,
* members of Portuguese Medical Association,
* authors of relevant scientific articles on medical education

Exclusion Criteria:

• Panelists who are not able to commit to all rounds of the modified Delphi process will be excluded.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Experts in Post-graduate medical education
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Consensus | 5 months
  The level of agreement for all statements achieving consensus from the expert panel consensus is predefined as ≥ 75% of the panel rating a given statement 4 or 5 value according to a Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Nuno L Fernandes, Principal Investigator — Centro Hospitalar do Baixo Vouga
Locations (1):
- Conselho Nacional do Internato Médico, Lisbon, Portugal

REFERENCES:
- See also: Research project website — https://epanf.pt/